CLINICAL TRIAL: NCT05511857
Title: Self-distancing and Pain: Can Different Thinking Strategies Affect the Perception of Short-lasting and Long-lasting, Persistent Pain?
Brief Title: Could Self-distancing Alter the Perception of Experimental Pain?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linnaeus University (Other)
Responsible Party: Principal Investigator, Helena Gunnarsson, Senior lecturer, Linnaeus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LinneausU
Record Dates: First submitted 2022-08-16; First posted 2022-08-23 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Pain, Experimental
Keywords: Pain
MeSH Terms: conditions — Pain | interventions — Osteogenesis, Distraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The effect of a self-distanced view on pain perception. (Experimental): The participant will exert self-distanced, third-person self-talk following a cue-card while induced with experimental pain.
  Interventions: Behavioral: Self-distancing, third-person self-talk.
- The effect of a self-immersed view on pain perception. (Experimental): The participant will exert self-immersed, first-person self-talk following a cue-card while induced with experimental pain.
  Interventions: Behavioral: Self-immersed, first-person self-talk.
- The effect of non-view, self-talk on pain perception. (Experimental): The participant will exert self-talk following a cue-card while induced with experimental pain.
  Interventions: Behavioral: Distraction
- Pain perception in induced, experimental pain. (No Intervention): Control group. This group will be induced with experimental pain, but will receive no specific task to exert.

INTERVENTIONS:
Behavioral: Self-distancing, third-person self-talk. — The participants will engage in self-distancing, third-person self-talk.
  Arms: The effect of a self-distanced view on pain perception.
Behavioral: Self-immersed, first-person self-talk. — The participants will engage in self-immersed, first-person self-talk.
  Arms: The effect of a self-immersed view on pain perception.
Behavioral: Distraction — The participants will engage in a distraction task.
  Arms: The effect of non-view, self-talk on pain perception.

SUMMARY:
Physical pain leads to a narrow, egocentric focus on the self, in the here and now, particularly when experienced at high intensity levels. When long-term pains are experienced, this narrow focus could be debilitating, since attention to the pain itself may increase its perceived intensity and it could increase negative emotional processes that further contribute to pain-related suffering. One way of overcoming this could be by adopting a more distant view of oneself and the pain, thereby making the pain more abstract. An established way of creating distance is by reflecting on the self, using one's own name and second or third-person singular pronouns, so called third-person self-talk. Earlier research has reported that a psychologically distant perspective could reduce emotional distress when reflecting on negative experiences, reduce feelings of anger after provocation and to lower blood pressure. Self-distancing should thus help people mentally reconstrue their pain experience and possibly make the pain signals less cognitively salient. In this experimental study, healthy participants will be induced with pain while performing different tasks.

DETAILED DESCRIPTION:
Physical pain leads to a narrow, egocentric focus on the self, in the here and now, particularly when experienced at high intensity levels. When long-term pain is experienced, this narrow focus could be debilitating, since attention to the pain itself may increase its perceived intensity and it could increase negative emotional processes that further contribute to pain-related suffering. One way of overcoming this could be by adopting a more distant view of oneself and the pain, thereby making the pain more abstract. An established way of creating distance is by reflecting on the self, using one's own name and second or third-person singular pronouns, so called third-person self-talk. Earlier research has reported that a psychologically distant perspective could reduce emotional distress when reflecting on negative experiences, reduce feelings of anger after provocation and lead to lower blood pressure. Self-distancing should thus help people mentally reconstrue their pain experience and possibly make the pain signals less cognitively salient.

In the first part of this study, which will be the first registered on ClinicalTrials.gov, we will experimentally induce pain in healthy participants (N = 292) with a cold pressor apparatus. The cold pressor apparatus holds a constant water temperature of 1 degree Celsius, which creates pain in the immersed hand. At the experimental test session, the participant will first be comfortably seated and receive information about the task and the experimental pain induction. They will be instructed to withhold their hand in the cold water for as long as possible, but when they feel that the pain becomes too intense they can choose to remove their hand. After that, a blood pressure measurement will be conducted. Directly after that, the participant will be instructed to put their hand in the cold water-bath (the cold pressor apparatus), and when they put their hand in the cold water a new blood pressure measurement will be conducted. A timer will be started to measure the time in seconds that the participant is able to keep their hand in the cold water. While their hand is in the cold water-bath, the participant will conduct one of the four different interventions (self-distanced, third-person self-talk following a cue-card; self-immersed, first-person self-talk following a cue-card; distraction intervention following a cue-card; no intervention (control)). When the participant removes their hand from the cold water-bath, the time in seconds will be noted and they will immediately be asked to estimate their pain on a Numerical Rating Scale. A short debriefing will conclude the session.

ELIGIBILITY:
Inclusion Criteria:

* No known disease affecting the nervous system.
* Swedish comprehension.
* Age over 18 years old.
* -

Exclusion Criteria

* Experiencing clinical pain at the test session.
* Known disease affecting the nervous system.
* Inadequate Swedish comprehension.
* Age under 18 years old.
* -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-06-09 (Estimated); Study Completion 2024-06-09 (Estimated)

PRIMARY OUTCOMES:
Pain tolerance | At the test session, the amount of time in seconds the participant withhold their hand in a cold water bath while engaging in self-talk will be measured. Data will be collected until study completion, approximately 1 year.
  The amount of time in seconds the participant can withhold their hand in the cold pressor test.
Pain intensity | The participant will be asked to estimate their pain from the hand (immersed in cold water) on the Numerical Rating Scale at the experimental test session. Data will be collected until study completion, approximately 1 year.
  The estimated experimental pain intensity on the Numerical Rating Scale. Minimum value of the Numerical Rating Scale is 0, which is equivalent with no pain. Maximum value of the Numerical Rating Scale is 10 which is equivalent of worst imaginable pain.
Pain-related fear | The participant will be asked to estimate their pain-related fear accompanying the pain they felt when the hand was immersed in cold water on the Numerical Rating Scale. Data will be collected until study completion, approximately 1 year.
  The estimated pain-related fear on the Numerical Rating Scale. Minimum value 0 and maximum value 10.
Change in blood pressure before and during pain induction. | The blood-pressure will be measured at the beginning of each test session and during the pain induction during each condition. Data will be collected until study completion, approximately 1 year..
  The difference score between the blood pressure before the pain induction and the blood pressure during the pain induction will be compared between the different groups. For example, the difference score between the blood pressure in the self-distanced, third-person self-talk condition will be compared to the difference score in the self-immersed, first-person self-talk condition.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Gunnarsson, PhD, Principal Investigator — Linnaeus University
Locations (1):
- Helena Gunnarsson, Vaxjo, Kronoberg County, Sweden

IPD SHARING:
Plan to Share IPD: No
No plan to share data.

REFERENCES:
- [Background] Ayduk, Ö., Kross, E. (2010). Analyzing Negative Experiences Without Ruminating: The Role of Self-Distancing in Enabling Adaptive Self-Reflection. Soc Personal Psychol Compass, 841-854. 10.1111/j.1751-9004.2010.00301.
- [Background] Loewenstein G. Out of control: visceral influences on behavior. Organ Behav Hum Decis Process. 1996;65(3):272-292.
- [Background] Mischkowski, D., Kross, E., Bushman, B.J. (2012). Flies on the wall are less aggressive: Self-distancing "in the heat of the moment" reduces aggressive thoughts, angry feelings, and aggressive behavior. J Exp Soc Psychol 48, 1187-1191.
- [Background] Orvell A, Vickers BD, Drake B, Verduyn P, Ayduk O, Moser J, Jonides J, Kross E. Does distanced Self-Talk Facilitate Emotion Regulation Across a Range of Emotionally Intense Experiences? Clin Psych Sci 2021; 9: 68-78.
- [Derived] Gunnarsson H, Agerstrom J. Pain From a Distance: Can Third-Person Self-Talk Mitigate Pain Sensitivity and Pain Related Distress During Experimentally Induced Pain? Psychol Rep. 2024 Aug 1:332941241269520. doi: 10.1177/00332941241269520. Online ahead of print. PMID 39091032